CLINICAL TRIAL: NCT03331406
Title: A Pilot Study of Physical Activity in Older Adults With Metastatic Gastrointestinal Cancer
Brief Title: Physical Activity In Gastrointestinal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jeffrey A. Meyerhardt, MD, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-350
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Gastrointestinal Cancer; Physical Activity
Keywords: Metastatic gastrointestinal cancer; Physical Activity
MeSH Terms: conditions — Gastrointestinal Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12-week physical activity program (Experimental): The physical activity program is of moderate intensity and consists of aerobic, strength, flexibility, and balance training with a target duration of 150 minutes per week.
  * At study start, participants will be provided with a pedometer to objectively monitor their aerobic activity, variable weight ankle weights and a medical journal to record physical activity.
  * Exercise Trainer --A exercise trainer will be assigned to design a physical activity program.
  Interventions: Other: Physical Activity Program

INTERVENTIONS:
Other: Physical Activity Program — 12-weeks in length, and includes moderate-intensity aerobic, strength, flexibility, and balance training.

SUMMARY:
This research study is evaluating the ability for people with metastatic gastrointestinal cancer to participate in a physical activity program.

DETAILED DESCRIPTION:
The physical activity program is 12-weeks in length, and includes moderate-intensity aerobic, strength, flexibility, and balance training.

* The goal of the aerobic training is to complete 150 minutes per week of brisk walking.
* The goals of the strength, flexibility, and balance training are to engage in these activities twice per week.

ELIGIBILITY:
Inclusion Criteria:

* Start of trial:

  * A three-month of strict inclusion criteria (Phase 1).
  * At the end of three-months, if at least six participants have not been accrued, inclusion criteria will be expanded for a second three-month recruitment phase (Phase 2).
  * At the end of six-months, an average of two patients per month has not been accrued, a further expand inclusion criteria (Phase 3).
* Phase 1 (most strict) Eligibility criteria include:

  * Voluntary, signed informed consent;
  * Diagnosis of histologically-confirmed esophageal, gastric, pancreatic, or colorectal that is metastatic or locally-advanced (unresectable);
  * First-line cytotoxic chemotherapy started within four-weeks of enrollment (patients can have reviewed prior adjuvant therapy if completed ≥6 months prior to start of first line chemotherapy for metastatic disease);
  * Age greater than 65 years;
  * Baseline weight-bearing physical activity less than 150 min∙wk-1 using the Paffenbarger physical activity questionnaire;
  * Eastern Cooperative Group Performance Status of 0, 1, or 2;
  * Self-reported ability to walk 400-meters (approximately one city block) without sitting, leaning, or the help of another person or walker;
  * Written physician approval;
  * Life expectancy >3 months;
  * English speaking.
* Phase 2 (less restrictive) Eligibility criteria will loosen:

  -- The minimum age from greater than 65, to greater than 55;
* Phase 3 (least restrictive) Eligibility criteria will add:

  -- The minimum age from greater than 55, to greater than 18.
* Exclusion Criteria

  * Known or suspected brain or other central nervous system metastases;
  * Uncontrolled cardiac or pulmonary disease;
  * Pregnant or breast feeding;
  * Any other condition that may impede testing of the study hypothesis, make it unsafe to engage in the physical activity program, or make the participant not available for end of study assessments (determined by the investigative team).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Rate of Accrual | 12 months
  Recruit 20 patients within 12 months
Number of participants that adhered to physical activity program | 12 Weeks
  Demonstrate that at least 50% of patients adhered to at least 50% of the prescribed physical activity program.

SECONDARY OUTCOMES:
Rate of Retention | 12 Weeks
  Proportion of participants who complete the study
Number of participants that complete assessment procedures | 12 Weeks
  Physical function testing and questionnaire collection
Number of participants with adverse events | 12 Weeks
  Falls, hospitalizations, and musculoskeletal injury

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Meyerhardt, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown JC, Brighton E, Campbell N, McCleary NJ, Abrams TA, Cleary JM, Enzinger PC, Ng K, Rubinson D, Wolpin BM, Yurgelun MB, Meyerhardt JA. Physical activity in older adults with metastatic gastrointestinal cancer: a pilot and feasibility study. BMJ Open Sport Exerc Med. 2022 May 30;8(2):e001353. doi: 10.1136/bmjsem-2022-001353. eCollection 2022. PMID 35722047